CLINICAL TRIAL: NCT05199714
Title: A Randomized, Controlled, Crossover Pilot Trial to Assess a Fully Automated, Dual-hormone (Insulin-and-pramlintide) Artificial Pancreas Without Carbohydrate Counting in Regulating Glucose Levels in Adults With Type 1 Diabetes
Brief Title: A Fully-closed Loop, Pramlintide and Insulin, Artificial Pancreas Clinical Trial for Adults With Type 1 Diabetes
Acronym: FCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Michael Tsoukas M.D., Principal Investigator, Assistant Professor, Endocrinology & Metabolism, McGill University Health Centre/Research Institute of the McGill University Health Centre, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8225
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas; Insulin; Pramlintide; Aspart; Fiasp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Aspart; Pancreas, Artificial; pramlintide

STUDY DESIGN:
Intervention Model Description: Randomized, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Fiasp-and-pramlintide fully automated system (8μg) (Experimental): Fiasp and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 8μg of pramlintide.
  Interventions: Drug: Fiasp; Device: Artificial Pancreas; Drug: Pramlintide
- Fiasp-alone with carbohydrate-matched boluses (Active Comparator): The Fiasp-alone intervention will have a 14 hour duration. During which, carbohydrate counting will inform insulin bolus doses based on insulin to carbohydrate ratios.
  Interventions: Drug: Fiasp
- Aspart-and-pramlintide fully automated system (10μg) (Experimental): Aspart and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 10μg of pramlintide.
  Interventions: Device: Artificial Pancreas; Drug: Pramlintide; Drug: Aspart
- Fiasp-and-pramlintide fully automated system (10μg) (Experimental): Fiasp and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 10μg of pramlintide.
  Interventions: Drug: Fiasp; Device: Artificial Pancreas; Drug: Pramlintide
- Aspart-and-pramlintide fully automated system (8μg) (Experimental): Aspart and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 8μg of pramlintide.
  Interventions: Device: Artificial Pancreas; Drug: Pramlintide; Drug: Aspart

INTERVENTIONS:
Drug: Fiasp — Fiasp Insulin delivered in a basal-bolus manner.
  Arms: Fiasp-alone with carbohydrate-matched boluses; Fiasp-and-pramlintide fully automated system (10μg); Fiasp-and-pramlintide fully automated system (8μg)
Device: Artificial Pancreas — Medtronic insulin pump, Dexcom G6 continuous glucose sensor, tablet running the Artificial Pancreas Algorithm.
  Arms: Aspart-and-pramlintide fully automated system (10μg); Aspart-and-pramlintide fully automated system (8μg); Fiasp-and-pramlintide fully automated system (10μg); Fiasp-and-pramlintide fully automated system (8μg)
Drug: Pramlintide — Pramlintide delivered in a basal-bolus manner.
  Arms: Aspart-and-pramlintide fully automated system (10μg); Aspart-and-pramlintide fully automated system (8μg); Fiasp-and-pramlintide fully automated system (10μg); Fiasp-and-pramlintide fully automated system (8μg)
Drug: Aspart — Aspart insulin delivered in a basal-bolus manner.
  Arms: Aspart-and-pramlintide fully automated system (10μg); Aspart-and-pramlintide fully automated system (8μg)

SUMMARY:
The investigators aim to assess the glycemic outcomes of a fully automated insulin-and-pramlintide artificial pancreas and a comparator insulin-alone artificial pancreas with carbohydrate matched boluses.

DETAILED DESCRIPTION:
The aim of this pilot study is to generate additional data of (i) a Fiasp-alone artificial pancreas with carbohydrate-matched boluses, compared to (ii) a Fiasp-plus-Pramlintide fully automated artificial pancreas with no meal announcement in an outpatient free-living setting. The study is not powered, nor aims to answer a scientific hypothesis related to the efficacy of the pramlintide and insulin closed-loop systems.

Design

The investigators will undertake a randomized crossover study to compare the following strategies:

1. Insulin-alone artificial pancreas with carbohydrate-matched boluses
2. Fiasp and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 8μg of pramlintide.
3. Fiasp and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 10μg of pramlintide.

   Each participant will be offered the opportunity to further participate in two optional additional arms:
4. Aspart and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 8μg of pramlintide.
5. Aspart and pramlintide artificial pancreas with no meal announcement. Ratio of 1 unit of insulin for 10μg of pramlintide.

Aspart is used in this optional arm as it is the slower-acting version of Fiasp and can therefore be used to draw reasonable comparisons. Further, Aspart is an FDA approved insulin which is commonly sold and prescribed in North America. Several co-formulations are being developed with insulin, pramlintide, and glucagon. Given the widespread adoption and use of Aspart, it makes this insulin a good candidate for use in co-formulations and an excellent option for transition to market, where they will impact many individuals living with diabetes.

Treatment period: Each intervention will last 14 hours. At-home run-ins, lasting two to four days, will occur prior to the pramlintide interventions. The interventions containing pramlintide with the same insulin will occur in sequence, one immediately after the other. The first pramlintide-and-Fiasp intervention will use a ratio of 8μg pramlintide/1unit of insulin and will be followed by the second pramlintide-and-Fiasp intervention the next day with a 10μg/1unit ratio. A similar schedule will be applied to the optional Aspart-and-pramlintide interventions. There will be a 2-29-day washout period between the Fiasp-and-pramlintide, Fiasp-alone, and Aspart-and-pramlintide interventions. Participants will be followed up remotely 1-2 days after the end of each intervention to ensure their washout period is going smoothly and will inquire about any adverse events. Remote contact can be performed via phone, email, text message or other reasonable communication channel. Participants will also be followed up remotely 1-2 days and 1-2 weeks after the end of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Females and males ≥ 18 years of age.
* Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Use of insulin pump therapy for at least 3 months.
* Effective birth-control use in individuals of childbearing potential. Individuals of child-bearing potential must agree to use a highly effective method of birth control.

Exclusion Criteria:

* Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2I (sodium-glucose transporter), GLP-1(glucagon-like peptide), Metformin, etc.).
* Current use of glucocorticoid medication (except low, stable does and inhaled steroids).
* Individuals with confirmed gastroparesis.
* Use of medication that alters gastrointestinal motility.
* Planned or ongoing pregnancy.
* Breastfeeding individuals.
* Severe hypoglycemia requiring hospitalization in the past three months.
* Severe diabetic ketoacidosis episode in the past three months.
* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event e.g., acute coronary syndrome or cardiac surgery.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Each participant's percentage of time glucose levels spent in the target range | 42 +/- 28 hours
  Time in target range (3.9-10.0 mmol/L).

SECONDARY OUTCOMES:
Each participant's percentage of time of glucose levels spent between 3.9 and 7.8 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's percentage of time of glucose levels spent below 3.9 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's percentage of time of glucose levels spent below 3.0 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's percentage of time of glucose levels spent above 10.0 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's percentage of time of glucose levels spent above 13.9 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's percentage of time of glucose levels spent above 16.7 mmol/L | 42 +/- 28 hours
  Glucose data will be collected from a glucose sensor and numerical glucose data will be analyzed as a function of time
Each participant's mean glucose levels | 42 +/- 28 hours
Each participant's standard deviation of glucose levels | 42 +/- 28 hours
Each participant's coefficient of variance of glucose levels | 42 +/- 28 hours
Total pramlintide delivery for each participant | 28 +/- 28 hours
Total insulin delivery for each participant | 42 +/- 28 hours
Total basal insulin delivery for each participant | 42 +/- 28 hours
Total bolus insulin delivery for each participant | 42 +/- 28 hours

OTHER OUTCOMES:
Safety Endpoints | 42 +/- 28 hours
  Adverse events including gastrointestinal symptoms (nausea, vomiting, diarrhea, bloating)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Center, Montreal, Quebec, Canada